CLINICAL TRIAL: NCT00287469
Title: A Phase II, Prospective, Randomized, Double-blind, Placebo Controlled, Field Efficacy Trial of a Candidate Hepatitis E Vaccine in Nepal.
Brief Title: A Safety and Efficacy Study of the Hepatitis E Vaccine in Nepal.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WRAIR 749; HSRRB A-9117.1; GSK 304558/003 (HEV-003); IND 7815 (Other: FDA)
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Results first posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Hepatitis
Keywords: Hepatitis E; clinical hepatitis; vaccine; efficacy; Nepal
MeSH Terms: conditions — Hepatitis; Hepatitis E

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 20mcg Recombinant HEV (Experimental): 20mcg of recombinant HEV antigen administered intramuscularly in the deltoid according to a 0, 1 and 6 month schedule
  Interventions: Biological: Hepatitis E vaccine, recombinant (Sar 56 kDa)
- Placebo (Placebo Comparator): PBS buffer placebo containing alum was administered intramuscularly in the deltoid according to a 0, 1 and 6 month schedule.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Hepatitis E vaccine, recombinant (Sar 56 kDa) — 20mcg or rhE Sar 56 kDa/dose of 0.5 mL, aluminium hydroxide (0.5 mg/dose) and phenoxyethanol (2.5 mg/dose)
  Arms: 20mcg Recombinant HEV
Other: Placebo — PBS buffer placebo containing alum
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if a hepatitis E vaccine is safe and able to prevent symptomatic liver disease due to the hepatitis E virus.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled with 2 study groups (vaccine and placebo). Three doses of the study vaccine are given according to a 0, 1, 6 month schedule. Vaccine efficacy will be assessed by maintaining active surveillance for clinical hepatitis every 2 weeks and hospital based surveillance for the full duration of the trial. Total planned study population is 2000 eligible subjects (1000 in the vaccine group and 1000 in the placebo group). Total vaccinated cohort for the analysis of reactogenicity is 200 (100 in the vaccine group and 100 in the placebo group).

Volunteers who enroll will be followed for evidence of symptomatic liver disease for approximately 2 years, and those who become ill will be admitted to hospital for care.

To evaluate safety, a randomly designated subset will be monitored for 7 days after each vaccination to solicit specific symptoms at the injection site and generally. Additionally, all adverse events will be collected for 30 days after each vaccine dose and all serious adverse events will be collected throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 18 years of age or older at the time of the first vaccination.
* Written or oral witnessed (if the subject was illiterate) informed consent obtained from the subject
* Free of obvious health problems as established by medical history before entering into the study
* If the subject was female, she must have a negative serum pregnancy test within 48 hours prior to each vaccination and must agree to avoid becoming pregnant during the course of vaccination and until 30 days after the last dose of vaccine.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune modifying drugs within six months of vaccination. For corticosteroids, this will mean prednisone, or equivalent, * 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Any chronic drug therapy to be continued during the study period with the exception of contraceptive agents, homeopathic remedies, vitamins, minerals and any other dietary supplements or other drug therapy at the discretion of the investigator.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine, excluding tetanus toxoid or rabies vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, as reported by the volunteer (testing for HIV will not be performed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrollment. Acute disease was defined as the presence of a moderate or severe illness with or without fever. All vaccines could be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., oral temperature < 38.0°C (100.4°F).
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by history.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant female.
* History of chronic alcohol consumption (defined as the consumption of the equivalent of 4 or more 12 ounce beers 4 or more times a week) and/or intravenous drug abuse.
* Antibodies to rHEV (* 20 WR U/mL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2001-07-09 (Actual); Primary Completion 2004-01-19 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mrigendra P Shrestha, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand; Robert M Scott, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Shree Birendra Hospital, Kathmandu, Nepal

REFERENCES:
- [Background] Worm HC, Schlauder GG, Brandstatter G. Hepatitis E and its emergence in non-endemic areas. Wien Klin Wochenschr. 2002 Aug 30;114(15-16):663-70. PMID 12602109
- [Background] Worm HC, van der Poel WH, Brandstatter G. Hepatitis E: an overview. Microbes Infect. 2002 May;4(6):657-66. doi: 10.1016/s1286-4579(02)01584-8. PMID 12048035
- [Background] Emerson SU, Purcell RH. Running like water--the omnipresence of hepatitis E. N Engl J Med. 2004 Dec 2;351(23):2367-8. doi: 10.1056/NEJMp048285. No abstract available. PMID 15575050
- [Background] Purcell RH. Hepatitis viruses: changing patterns of human disease. Proc Natl Acad Sci U S A. 1994 Mar 29;91(7):2401-6. doi: 10.1073/pnas.91.7.2401. PMID 8146130
- [Background] Worm HC, Wirnsberger G. Hepatitis E vaccines: progress and prospects. Drugs. 2004;64(14):1517-31. doi: 10.2165/00003495-200464140-00002. PMID 15233590
- [Derived] Shrestha MP, Scott RM, Joshi DM, Mammen MP Jr, Thapa GB, Thapa N, Myint KS, Fourneau M, Kuschner RA, Shrestha SK, David MP, Seriwatana J, Vaughn DW, Safary A, Endy TP, Innis BL. Safety and efficacy of a recombinant hepatitis E vaccine. N Engl J Med. 2007 Mar 1;356(9):895-903. doi: 10.1056/NEJMoa061847. PMID 17329696

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2000 subject were recruited by Royal Nepalese Army investigators at the Shree Birendra Hospital, Kathmandu from a well characterized population of Royal Nepalese Army military personnel stationed in the Kathmandu Valley and their family members and up to 5 US citizens residing in the Nepal.
Period: Overall Study
Arm/Group | Placebo | 20mcg Recombinant HEV
Started | 1000 | 1000
Completed | 780 | 786
Not Completed | 220 | 214
Not completed — serious adverse event | 1 | 6
Not completed — Adverse Event | 1 | 1
Not completed — moved from area | 144 | 138
Not completed — Lost to Follow-up | 74 | 69

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 20mcg Recombinant HEV | Total
Number analyzed (Participants) | 1000 | 1000 | 2000
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Male and Female participants add up to the total number for each group: Placebo (1000) and 20mcg Recombinant HEV (1000).
  Years
    Female: number analyzed (Participants) | 4 | 4 | 8
    Female | 31.3 (12.69) | 28.0 (8.29) | 29.6 (10.07)
    Male: number analyzed (Participants) | 996 | 996 | 1992
    Male | 25.1 (6.12) | 25.2 (6.34) | 25.2 (6.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 996 | 996 | 1992
Region of Enrollment [Number; unit: participants]
  Nepal | 1000 | 1000 | 2000

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants of Definite Hepatitis E by Category and Immunological Markers (Anti HEV) During the Follow-up Period
Description: Percent of participants of definite hepatitis E by category and immunological markers (anti HEV) during the follow-up period.
  * Illness for at least 3 days comprised of at least 3 of the following symptoms: fatigue, loss of appetite, abdominal discomfort, right upper quadrant pain, nausea, vomiting
  * Peak of Alanine Aminotransferase (ALT) greater then 2.5 times the upper limit of normal (2.5 x 42 =105)
  * Percent of Participants = n x 100 / N
Time Frame: 14 days after dose 3 at 6 months
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | 20mcg Recombinant HEV | Placebo
Number analyzed (Participants) | 1000 | 1000
Percent of Participants
  Jaundice; IgM ≥ 100 WR U/mL | 0.0 [0.0 to 0.4] | 6.9 [5.3 to 8.8]
  Jaundice; total lg ≥ 2500 WR U/mL | 0.3 [0.1 to 1.0] | 0.1 [0.0 to 0.6]
  Jaundice; IgM≥100 WR U/mL or total lg≥2500 WR U/mL | 0.3 [0.1 to 1.0] | 7.0 [5.4 to 8.9]
  Illness; IgM ≥ 100 WR U/mL | 0.0 [0.0 to 0.4] | 0.3 [0.1 to 1.0]
  Illness; total lg ≥ 2500 WR U/mL | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Illness; IgM≥100 WR U/mL or total lg≥2500 WR U/mL | 0.0 [0.0 to 0.4] | 0.3 [0.1 to 1.0]
  Jaun/Ill; IgM≥100 WR U/mL or total lg≥2500 WR U/mL | 0.3 [0.1 to 1.0] | 7.4 [5.7 to 9.3]

2. Secondary Outcome: Percent of Participants of Definite Hepatitis E Disease by Category During the Follow-up Period
Description: Percent of participants of definite hepatitis E and vaccine efficacy by category during the follow-up period
  * Illness for at least 3 days comprised of at least 3 of the following symptoms: fatigue, loss of appetite, abdominal discomfort, right upper quadrant pain, nausea, vomiting
  * Peak of Alanine Aminotransferase (ALT) greater then 2.5 times the upper limit of normal (2.5 x 42 =105)
  * Percent of participants = n x 100 / N
Time Frame: 14 days after dose 2 until 14 days after dose 3
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | 20mcg Recombinant HEV | Placebo
Number analyzed (Participants) | 1000 | 1000
Percent of Participants
  Jaundice; IgM ≥ 100 WR U/ml | 0.1 [0.0 to 0.6] | 0.8 [0.4 to 1.6]
  Jaundice; total Ig ≥ 2500 WR U/ml | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Jaundice; IgM≥100 WR U/mL or total lg≥2500 WR U/mL | 0.1 [0.0 to 0.6] | 0.8 [0.4 to 1.6]
  Illness; ImG ≥ 100 WR U/ml | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Illness; total Ig ≥ 2500 WR U/ml | 0.0 [0.0 to 0.4] | 0.0 [0.0 to 0.4]
  Jaun/Ill; IgM≥100 WR U/mL or total lg≥2500 WR U/mL | 0.1 [0.0 to 0.6] | 0.8 [0.4 to 1.6]

3. Secondary Outcome: Number of Suspected, Definite, Probable and Not Confirmed Hepatitis E Disease Cases
Description: Number of suspected, definite, probable and not confirmed hepatitis E disease cases during surveillance period
Time Frame: before dose 1 thru 14 days after dose 3
Measure: Number; unit: Number of Hepatitis E Cases
Arm/Group | Placebo | 20mcg Recombinant HEV
Number analyzed (Participants) | 1000 | 1000
Number of Hepatitis E Cases
  Any acute hep cases: before dose 1 | 0 | 1
  Any hep cases: within 14 days after dose 1 | 1 | 3
  Any hep cases: between 14 days after dose 1 and 2 | 5 | 2
  Any hep cases: within 14 days after dose 2 | 0 | 0
  Any hep cases: between 14 days after dose 2 and 3 | 7 | 4
  Any hep cases: within 14 days after dose 3 | 1 | 0
  Any hep cases: from 14 days after dose 3 | 78 | 9
  Any hep cases: Total | 92 | 19
  Definite hepE cases: before dose 1 | 0 | 0
  Definite hepE cases: within 14 days after dose 1 | 1 | 3
  Definite hepE cases: btwn 14dys after dose 1 and 2 | 3 | 2
  Definite hepE cases: within 14 days after dose 2 | 0 | 0
  Definite hepE cases: btwn 14dys after dose 2 and 3 | 7 | 1
  Definite hepE cases: within 14 days after dose 3 | 1 | 0
  Definite hepE cases: from 14 days after dose 3 | 66 | 3
  Definate hepE cases: Total | 78 | 9
  Probable hepE cases | 0 | 0
  Not confirmed hepE: before dose 1 | 0 | 1
  Not confirmed hepE: within 14 days after dose 1 | 0 | 0
  Not confirmed hepE: btwn 14dys after dose 1 and 2 | 2 | 0
  Not confirmed hepE: within 14 days after dose 2 | 0 | 0
  Not confirmed hepE: btwn 14dys after dose 2 and 3 | 0 | 3
  Not confirmed hepE: within 14 days after dose 3 | 0 | 0
  Not confirmed hepE: from 14 days after dose 3 | 12 | 6
  Not confirmed hepE: total | 14 | 10

ADVERSE EVENTS:
Time Frame: Within 31 days (days 0-30) post-vaccination
Arm/Group | Placebo | 20mcg Recombinant HEV
All-Cause Mortality (participants affected / at risk) | 1/1000 | 6/1000
Serious Adverse Events (participants affected / at risk) | 200/1000 | 143/1000
Other Adverse Events (participants affected / at risk) | 226/1000 | 229/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1000) | 20mcg Recombinant HEV (N=1000)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Gilbert's syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Accidental death (General disorders) | 1 (1) | 0 (0)
Carcadian rhythm sleep disorder (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 5 (5)
Gravitational oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 6 (6) | 1 (1)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 2 (2)
Jaundice hepatocellular (Hepatobiliary disorders) | 5 (5) | 2 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Amoebiasis (Infections and infestations) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 3 (3)
Ascariass (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cestode infection (Infections and infestations) | 1 (1) | 0 (0)
Dermatitis infection (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 3 (3) | 1 (1)
Encephalitis japanese b (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Giardiasis (Infections and infestations) | 3 (3) | 6 (6)
Hepatitis E (Infections and infestations) | 81 (81) | 10 (10)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Hookworm infection (Infections and infestations) | 4 (4) | 3 (3)
Hymenolepiasis (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 3 (3) | 1 (1)
Leptospirosis (Infections and infestations) | 12 (12) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Malaria (Infections and infestations) | 3 (3) | 1 (1)
Measles (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 2 (2) | 1 (1)
Neurocysticercosis (Infections and infestations) | 1 (1) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media chronic (Infections and infestations) | 0 (0) | 2 (2)
Paratyphoid fever (Infections and infestations) | 7 (7) | 8 (8)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 0 (0)
Respiratory tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 3 (3) | 7 (7)
Scrub typhus (Infections and infestations) | 3 (3) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Tonsilitis (Infections and infestations) | 3 (3) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 24 (24) | 30 (30)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 6 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 9 (9) | 5 (5)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blast injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 3 (3) | 9 (9)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Polytraumatism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 5 (5)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Costochandritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebrial disc protrution (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatic fever (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroilitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 4 (4)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Phimosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Nasal septum (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Anal fistula excision (Surgical and medical procedures) | 1 (1) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 2 (2)
Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Vasectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Wound haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1000) | 20mcg Recombinant HEV (N=1000)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 15 (15)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 22 (22) | 22 (22)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 9 (9)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pericoronitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 5 (5) | 6 (6)
Chest pain (General disorders) | 3 (3) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (3)
Feeling of body temperature change (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Injection site anaesthesia (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 5 (5) | 6 (6)
Pyrexia (General disorders) | 31 (31) | 29 (29)
Jaundice hepatocellular (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 3 (3) | 3 (3)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Acute tonsillitis (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
Ascariasis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Dermatitis infected (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Dysentery (Infections and infestations) | 2 (2) | 3 (3)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis japanese b (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 2 (2)
Furuncle (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1) | 3 (3)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1)
Helminthic infection (Infections and infestations) | 1 (1) | 2 (2)
Hepatitis e (Infections and infestations) | 3 (3) | 4 (4)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 2 (2) | 1 (1)
Leptospirosis (Infections and infestations) | 3 (3) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (20) | 22 (22)
Otitis media chronic (Infections and infestations) | 0 (0) | 2 (2)
Paratyphoid fever (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Scrub typhus (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 11 (11) | 8 (8)
Typhoid fever (Infections and infestations) | 6 (6) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 9 (9)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 5 (5) | 4 (4)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heat exhaustion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Post procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 10 (10) | 4 (4)
Headache (Nervous system disorders) | 43 (43) | 36 (36)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 4 (4)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Neophrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 0 (0) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 2 (2)
Vasectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Wart excision (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No